CLINICAL TRIAL: NCT05369130
Title: Characterising the Phenotype for Persistent Postoperative Pain Following Repair of the Thoraco-abdominal Aorta
Brief Title: Investigate and Predict Aortic & Thoracic Surgery Persistenet Postsurgical Pain
Acronym: ImPARTonPPP
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 303825
Record Dates: First submitted 2022-02-22; First posted 2022-05-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Persistent Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Acellular CSF and Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Develop Persistent Postsurgical Pain: Pain present 3 months post-op related to the surgical operation
- Absence of Persistent Postsurgical Pain: Resolution of post-operative pain within the first three months of the operation

SUMMARY:
This is an observational clinical study aiming to further the wider understanding of patients who develop persistent pain after Thoracoabdominal Aorta surgery, a surgical cohort who are disproportionately affected. This will be undertaken through a prospective biopsychosocial characterisation of the phenotype of patients undergoing this operation.

Increasing numbers of patients are undergoing surgery on the chest for treatment of heart or lung cancer disease. Over the last twenty years, the medical community has become increasingly aware of the long-term effect of this surgery in producing persistent pain, approximately half of all survivors are still in pain around their surgical incision at three months postoperatively and beyond. There is currently no accepted method for preventing this phenomenon.

The nervous system mechanisms for the development of persistent pain after surgery are unclear. Some studies suggest it may involve the patient's ability to dampen down pain signals travelling from the incision site to the brain.

Humans have an in-built system that produces opiates as well as other pain-relieving molecules in response to injury, e.g. surgery. However, this response varies hugely from person to person and may even be impacted by the psychological state of the individual at the time of surgery. Some of these pain modulating mechanisms can be measured before and after surgery in patients using sensory testing, a robust and established objective method to assess patients'.

Identifying patients who are most at risk of a persistent pain state will allow both academics and clinicians to investigate and better target appropriate treatments.

Undertaking these longitudinal observational assessments will facilitate an improved mechanistic insight of the transition from acute to pathological pain, with the ultimate goal of improving outcomes for patients'.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years of age) undergoing elective repair of the thoraco-abdominal aorta. Able to adequately understand and respond to verbal instructions

Exclusion Criteria:

* Unwilling or unable to give consent, Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults Undergoing Elective Repair of the thoraco-abdominal aorta
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Characterise the sensory phenotype of Persistent Postsurgical Pain following Thoracoabdominal Aortic Surgery with Quantitative Sensory Testing as a change measure. | 3 Years
  Quantitative Sensory Tests (Pre-op, Early Post-operative Period, > 3 months Post-op)
Characterise the Pain Intensity as a change measure following Thoracoabdominal Aortic Surgery | 3 years
  Pain Intensity as measured by Visual Analogue Score (Pre-Op, Pre discharge, after three months post-op)
Characterise the Pain Intensity as a change measure following Thoracoabdominal Aortic Surgery | 3 years
  Pain Intensity as measured by Numerical Rating Score (Pre-Op, Throughout the peri-op period and till 2 years post-op)
Characterise the analgesia requirements as a change measure following Thoracoabdominal Aortic Surgery | 3 years
  Analgesic requirements as measured by oral morphine equivalents (Pre-Op, Throughout the peri-op period and till 2 years post-op)
Characterise the analgesia requirements as a change measure following Thoracoabdominal Aortic Surgery | 3 years
  Non-opioid analgesic prescriptions (Pre-Op, Throughout the peri-op period and till 2 years post-op)
Characterise the presence of neuropathic sensory phenotype of patients undergoing Thoracoabdominal Aortic Surgery pre-op, post-op and > 3 months post-op. | 3 years
  Neuropathic Pain as defined by Douleur Neuropathique 4 (DN4) (Pre-Op, > 3 months Post-op and till 2 years post-op)
Characterise the presence of neuropathic sensory phenotype of patients undergoing Thoracoabdominal Aortic Surgery pre-op, post-op and > 3 months post-op. | 3 years
  Neuropathic Pain as defined by Self Reported Leeds Assessment of Neuropathic Symptoms and Signs (SLANSS) (Pre-Op, > 3 months Post-op and till 2 years post-op)
Characterise the change in biochemical phenotype pre-op and in the early post-op period following Thoracoabdominal Aortic Surgery and define significant differences between those with and without persistent post surgical pain | 3 Years
  Multi regression analysis of CSF composition.
Characterise the change in biochemical phenotype pre-op and in the early post-op period following Thoracoabdominal Aortic Surgery and define significant differences between those with and without persistent post surgical pain | 1 Week
  Multi regression analysis of blood composition.
Identify Predictors of Persistent Postsurgical Pain following Thoracoabdominal Aorta surgery | 3 years
  Determine if a composite biomarker or non response to conditioned pain modulation is a biomarker for development of persistent post-surgical pain and whether these are associated with biochemical differences through a bioinformatic data analysis approach.

SECONDARY OUTCOMES:
Determine the influence of baseline psychological and social profiles on postoperative pain outcomes. | 3 years
  Measured with Pain Catastrophising Scale (PCS) (Pre-Op, > 3 months Post-op)
Determine the influence of baseline psychological and social profiles on postoperative pain outcomes. | 3 years
  Pain Anxiety Symptom Scale PASS20 as a change measure over time (Pre-Op, > 3 months Post-op)
Determine the influence of baseline psychological and social profiles on postoperative pain outcomes. | 3 years
  Patient-Reported Outcomes Measurement Information System PROMIS: Fatigue and Sleep, depression and Anxiety as a change measure over time. (Pre-Op, > 3 months Post-op)
Describe the impact of Persistent Post Surgical Pain on Quality of Life | 3 years
  Changes in EuroQual 5 Dimensions EQ5D. (Pre-Op, > 3 months Post-op and till 2 years post-op)

CONTACTS AND LOCATIONS:
Overall Officials: Sibtain Anwar, MBBS MA PhD, Study Chair — Barts Health NHS Trust & Queen Mary University of London
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data will be made available